CLINICAL TRIAL: NCT01690494
Title: Protect and Connect: Couple HIV Prevention for Drug Involved Male Offenders, An Effectiveness Trial
Brief Title: Protect and Connect: Couple HIV Prevention for Drug Involved Male Offenders
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nabila El-Bassel, PhD, Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAK0206; 1R01DA033168-01A1 (NIH)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Sexually Transmitted Diseases; Unsafe Sex; Substance-Related Disorders
Keywords: STI; sexually transmitted infection; HIV; criminal justice; probation; couples; drug use
MeSH Terms: conditions — Sexually Transmitted Diseases; Unsafe Sex; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT + TAU (Experimental): 4-session PACT delivered to both partners together + standard treatment of care services (TAU) delivered to the male participant
  Interventions: Behavioral: PACT; Behavioral: TAU
- TAU (Active Comparator): TAU control condition delivered to the male participant
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: PACT — Couple-based behavioral HIV/STI preventive intervention
  Arms: PACT + TAU
Behavioral: TAU — Standard treatment of care services provided to male offenders by the Criminal Court, Community Court or probation sites

SUMMARY:
This study is a randomized controlled trial (RCT) that will rigorously evaluate the implementation, effectiveness and cost-effectiveness of a couple-based integrated human immunodeficiency virus (HIV) and drug abuse prevention intervention (Connect II) with drug-involved male offenders charged with misdemeanors and their primary female sexual partners, implemented by frontline providers in Criminal Court, Community Court or probation (CCP) sites in NYC, compared to CCP standard treatment of care services (TAU). The primary outcomes are to reduce sexually transmitted infections (STIs) and increase condom use.

DETAILED DESCRIPTION:
HIV/acquired immune deficiency syndrome (AIDS) and criminal justice involvement are critical intersecting public health issues for drug-involved men. Low income, Black and Hispanic men especially bear the burden of the HIV epidemic and are over-represented in the U.S. criminal justice system. Recent Centers for Disease Control and Prevention (CDC) surveillance data suggest that the health disparity in HIV rates is actually increasing for Black men: current estimates suggest 1 in 16 Black men in the U.S. will be infected with HIV in their life time. These HIV/STI transmission risks are fueled by high rates of poverty, incarceration, unemployment, and lack of access to health care and prevention services. The proposed study thus targets an underserved population at the epicenter of the epidemic in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Couples
* Both partners are aged 18 or older
* Identify each other as their primary sexual partner of opposite sex
* Relationship has existed at least 3 months
* At least one partner reports having unprotected vaginal or anal intercourse with the other partner in the past 90 days
* At least one partner reports exposure to an outside HIV risk in the past year
* Male partner reports and is verified by court records of being charged with a misdemeanor
* Male partner is currently under court supervision or probation

Exclusion Criteria:

* Either partner shows evidence of significant psychiatric or could impairment as confirmed by the MacArthur Competence Assessment Tool during the screening eligibility interview.
* Either partner reports severe physical or sexual violence perpetrated by the other partner in the past year as measured on the Revised Conflict Tactics Scale
* Either partner is unable to commit to participate in the study through to completion
* Either partner reports that the couple is planning a pregnancy within the next 12 months
* Either partner is not fluent in English as determined during Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in biologically confirmed sexually transmitted infections | Baseline and up to 12 months post intervention
Change in proportion of unprotected sexual acts | Baseline and up to 12 months post intervention

SECONDARY OUTCOMES:
Change in drug use | Baseline and up to 12 months post intervention
Change in utilization of drug treatment | Baseline and up to 12 months post intervention
Change in recidivism | Up to 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nabila El-Bassel, DSW, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El-Bassel N, Gilbert L, Wu E, Witte SS, Chang M, Hill J, Remien RH. Couple-based HIV prevention for low-income drug users from New York City: a randomized controlled trial to reduce dual risks. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):198-206. doi: 10.1097/QAI.0b013e318229eab1. PMID 21725249
- [Derived] Wimberly AS, Rose R, Levin K, Goddard-Eckrich D, Gilbert L, Wu E, Dasgupta A, Hunt T, Henry BF, El-Bassel N. Traumatic Life Events and Stressors: Associations With Substance Use Problems of Men Under Community Supervision. J Correct Health Care. 2023 Jun;29(3):190-197. doi: 10.1089/jchc.21.12.0137. Epub 2023 Apr 28. PMID 37116052
- [Derived] El-Bassel N, Gilbert L, Goddard-Eckrich D, Chang M, Wu E, Goodwin S, Tibbetts R, Almonte-Weston M, Hunt T. Effectiveness of a Couple-Based HIV and Sexually Transmitted Infection Prevention Intervention for Men in Community Supervision Programs and Their Female Sexual Partners: A Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e191139. doi: 10.1001/jamanetworkopen.2019.1139. PMID 30924895